CLINICAL TRIAL: NCT00018265
Title: Oxygen Kinetics, Mobility Task Performance, and Task Training in Older Adults
Brief Title: Fitness and Daily Function in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AGCG-003-99S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Cardiovascular Disease
Keywords: Rehabilitation; exercise test; aging
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tai Ji

INTERVENTIONS:
Behavioral: Task specific endurance training
Behavioral: Tai Chi

SUMMARY:
The purpose of this study is to examine the impact of aerobic fitness on the ability of able and disabled older adults to perform daily functional activities. Subjects are tested in their oxygen use patterns as they perform a series of functional tasks (such as walking on stairs) and following a 24-week training program focused on improving the ability to perform daily tasks likely requiring aerobic fitness (such as walking on stairs).

ELIGIBILITY:
Both healthy and self-reported mobility-impaired older adults

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140
Dates: Start 1999-10; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Donald Dengel
Locations (1):
- Ann Arbor Healthcare System, Ann Arbor, Michigan, United States